CLINICAL TRIAL: NCT04805359
Title: Effect of Hypoxia Exercise on Erythrocyte Aggregability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jong-Shyan Wang, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200903510B0
Record Dates: First submitted 2021-02-25; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Hypoxia; Training
Keywords: Erythrocyte; Aggregation
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normoxic exercise (NE) (Experimental): The subjects were trained on a bicycle ergometer at 60% of maximal work-rate (60%Wmax) under 21%O2 in air (NE) for 30 minutes per day, 5 days per week for 6 weeks
  Interventions: Behavioral: Normoxic exercise
- Hypoxic exercise (HE) (Experimental): The subjects were trained on a bicycle ergometer at 60% of maximal work-rate (60%Wmax) under 15%O2 in air (HE) for 30 minutes per day, 5 days per week for 6 weeks
  Interventions: Behavioral: Hypoxic exercise
- Normoxic control (No Intervention): Without any exercise training

INTERVENTIONS:
Behavioral: Normoxic exercise — Trained on a bicycle ergometer at 60% of maximal work-rate (60%Wmax)for 30 minutes per day, 5 days per week for 6 weeks
  Arms: Normoxic exercise (NE)
Behavioral: Hypoxic exercise — Trained on a bicycle ergometer at 60% of maximal work-rate (60%Wmax)for 30 minutes per day, 5 days per week for 6 weeks
  Arms: Hypoxic exercise (HE)

SUMMARY:
Pathological erythrocyte aggregation reduces capillary perfusion and oxygen transfer to tissue. The aggregation is determined by opposing forces, the repulsive force between cells, cell-to-cell adhesion induced by plasma fibrinogen, and the disaggregating shear force generated by blood flow. The investigators investigate how hypoxic exercise affects intrinsic/extrinsic factors of aggregation. Sixty sedentary males were randomly assigned into either hypoxic (HE; FiO2=15%, n=20) or normoxic (NE; FiO2=21%, n=20) training groups for 30 min·d-1, 5 d·wk-1 for 6 weeks at 60% of maximum work rate or to a control group (CTL; n=20). A hypoxia exercise test (HET, FiO2=12%) was performed before and after the intervention. The erythrocyte aggregation, binding affinity of fibrinogen and membrane biomarkers were determined by an ektacytometry and flow cytometry, respectively.

DETAILED DESCRIPTION:
The aim of this study is to clarify the effects of exercise training with and without hypoxia on the erythrocyte aggregation, further providing a feasible strategy for developing an appropriate exercise regimen that improves cardiopulmonary fitness and minimizes the risk of hemorheological disorders. This study evaluated the distinct effects of hypoxic exercise training (HE) and normaxia exercise training (NE) for 6 weeks on the following issue: (1) intrinsic/extrinsic erythrocyte aggregation, (2) binding affinity of fibrinogen to erythrocyte, (3) erythrocyte turnover rate and (4) characteristic of mature erythrocytes in blood, under hypoxic exercise test (HET) (100W under air 12% O2 condition) in healthy sedentary men.

ELIGIBILITY:
Inclusion Criteria:

* Having a sedentary lifestyle (without regular exercise, exercise frequency ≤ once weekly, duration < 20 min).

Exclusion Criteria:

* Exposed to high altitudes (> 3000 m) for at least 1 year.
* Smoker
* Taking medications or vitamins
* Having any cardiopulmonary/hematological risk.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07-05 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-06-30 (Actual)

PRIMARY OUTCOMES:
Total Erythrocyte Aggregation | 8 weeks
  The total erythrocyte aggregation was determined by using Microfluidic Ektacytometer (Rheoscan-AnD 300, RheoMeditech, Seoul, Korea).

SECONDARY OUTCOMES:
Cardiopulmonary capacity | 8 weeks
  To assess cardiopulmonary capacity, the cardiopulmonary exercise test (CPET) on a cycle ergometer was performed 4 days before and after the intervention. All subjects underwent exercise with a mask to measured oxygen consumption (VO2) breath by breath using a computer-based system (Master Screen CPX, Cardinal-health Germany). After 5-min baseline resting period records, a 2-min warm-up period (60 rpm, unloaded pedaling) was started and followed by an incremental work (30 W elevation for each 3-minute) until exhaustion (i.e., progressive exercise to maximal O2 consumption, VO2max).
The affinity between erythrocyte and fibrinogen | 8 weeks
  1. The erythrocyte suspension (1×10^6 cells/μl) was incubated with fibrinogen (400 mM) and anti-fibrinogen-FITC monoclonal antibody (1:500, Cedarlane) in the dark for 30 min at RT.
  2. After the staining is completed, add 1μl suspension into 100μl medium solution, then rotate the sample on a Viscometer (Brookfield) at different rates (0, 50, 100, 200, 400, 800 rpm) for 1 min at 37°C in the dark.
  3. The mean fluorescence intensity (MFI) obtained from 50,000 erythrocytes was measured by FACSCalibur (Becton Dickinson, New Jersey, USA).
Senescence-Related Molecules on Erythrocyte | 8 weeks
  Erythrocyte suspensions (1x10^6 cells /µl) were incubated with monoclonal anti- CD147(eBioscience) and anti-CD47(BioLegend) that were conjugated with FITC in the dark for 30 min at 37°C. The MFI obtained from 50,000 erythrocytes was measured by using FACSCalibur.
Adhesion-Related Molecules on Erythrocyte | 8 weeks
  Erythrocyte suspensions (1x10^6 cells /µl) were incubated with monoclonal anti-CD49d (eBioscience) and anti- CD36(BioLegend) that were conjugated with FITC in the dark for 30 min at 37°C. The MFI obtained from 50,000 erythrocytes was measured by using FACSCalibur.
The influences of fibrinogen to erythrocytes | 8 weeks
  1. The hematocrit (Hct) of erythrocyte sample was adjusted to 40% to eliminate the effect of dehydration after exercise.
  2. The adjusted sample was pre-treated with 400 mM fibrinogen for 30 min.
  3. The erythrocyte aggregation was determined by using Microfluidic Ektacytometer (Rheoscan-AnD 300, RheoMeditech, Seoul, Korea).
The influences of the intrinsic factor to erythrocytes | 8 weeks
  1. The hematocrit (Hct) of erythrocyte sample was adjusted to 40% to eliminate the effect of dehydration after exercise.
  2. The adjusted sample was pre-treated with 10 mM Dextran for 30 min.
  3. The erythrocyte aggregation was determined by using Microfluidic Ektacytometer (Rheoscan-AnD 300, RheoMeditech, Seoul, Korea).
The influences of the extrinsic factor to erythrocytes | 8 weeks
  1. The hematocrit (Hct) of erythrocyte sample was adjusted to 40% to eliminate the effect of dehydration after exercise.
  2. For excluding the effect of changed plasma composition, the erythrocyte sample was added into the platelet-poor-plasma (PPP) collected before the hypoxia exercise test.
  3. The erythrocyte aggregation was determined by using Microfluidic Ektacytometer (Rheoscan-AnD 300, RheoMeditech, Seoul, Korea).

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Shyan Wang, PhD, Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No